CLINICAL TRIAL: NCT02603848
Title: Assessing the Effectiveness of Ibuprofen Compared to Morphine as a Pediatric Postoperative Pain Management Tool Following Inguinal Surgery (AIMS)
Brief Title: Ibuprofen Compared to Morphine as a Pediatric Postoperative Pain Management Tool Following Inguinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ibuprofen vs. Morphine
Record Dates: First submitted 2015-09-25; First posted 2015-11-13 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Inguinal Surgery
Keywords: Inguinal surgery; Hernia Repair; Orchidopexy; Hydrocele; Pediatric; Post-operative pain; Morphine sulfate; Ibuprofen
MeSH Terms: conditions — Testicular Hydrocele; Pain, Postoperative | interventions — Ibuprofen; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen suspension (Experimental): Ibuprofen suspension (Advil) will be administered orally at a dose of 10mg/kg every 6 hours for 72 hours post-surgery.
  Interventions: Drug: Ibuprofen
- Morphine Sulfate suspension (Active Comparator): Morphine sulfate suspension will be administered orally at a dose of 0.02 - 0.04 mg/kg every 6 hours for 72 hours post-surgery.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ibuprofen — (10mg/kg; maximum 600 mg) every six hours as needed
  Other Names: Advil
  Arms: Ibuprofen suspension
Drug: Morphine — 0.2 mg/ kg morphine suspension (maximum 10mg) every four hours as needed
  Other Names: Morphine sulfate
  Arms: Morphine Sulfate suspension

SUMMARY:
Morphine is now the most commonly used opioid in children for pain management even though the safety of morphine use in children is a primary concern for parents as it is perceived to have more associated risks. Ibuprofen and other Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) have also been shown to be effective for the management of postoperative pain with fewer associated adverse effects. However, there have been concerns that utilization of ibuprofen alone may lead to inadequate pain management. Evidence of whether ibuprofen is equally effective as morphine for postoperative pain control in pediatric inguinal surgery is lacking and needs to be further explored as a measure to potentially reduce opioid exposure in children. To determine which drug is more effective for relieving post-operative pain, this trial will compare the effectiveness of ibuprofen and morphine at reducing post-operative pain, and the amount of analgesic use required post-surgery.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the efficacy of ibuprofen in reducing postoperative pain in children recovering from inguinal surgery when compared to morphine. Thus, if stated as a research question, the problem to be addressed is: in children (10 months-5 years) who have recently undergone inguinal surgery, is ibuprofen, when administered postoperatively, no less effective in reducing postoperative pain compared to morphine? Inguinal surgical procedures (unilateral hernia/ hydrocele repair and unilateral orchidopexy) will be carried out under standardized analgesic administration. Anesthesia will be delivered to all participants via inhalation induction with air/nitrous oxide and sevoflurane, intravenous supplementation with propofol and/or fentanyl 1 to 2 mcg/kg, antiemetic prophylaxis with dexamethasone 150 mcg/kg and ondansetron 50 mcg/kg, acetaminophen suppository 40 mg/kg, and morphine intravenous 50-100 mcg/kg. Regional block with local infiltration of 0.25 % of plain bupivacaine will be performed around the vicinity of the ileoinguinal nerve. This anesthesia protocol has been approved by a consensus meeting with the Pediatric Anesthesia Group at McMaster University and will be employed consistently in all cases in this study. Deviations to this practice will lead to study exclusion.

Postoperatively, the control group will receive standardized 0.2 mg/ kg morphine syrup (maximum 10mg) every four hours as needed, while the intervention group will receive Ibuprofen suspension (10mg/kg; maximum 600 mg) every six hours as needed for 48 hours post hospital discharge. Tylenol (15mg/kg) can be administered in either group at parental discretion every four hours as needed and will be recorded in a standardized medication log provided to all parents.

Parents will be told to follow the instructions on the package of prefilled syringes (i.e. to give the medication every 4 hours or 6 hours as needed) by the healthcare practitioner who is discharging the patient from the hospital. Parents and will not be told which medication their child is receiving in order to maintain blinding. All dosage information will be kept and maintained by the research pharmacy staff. Parents will be provided medication information through the use of a standardized script and hand out available in both English and French which will encompass potential side effects of both trial medications.

The duration of the treatment period will be following hospital discharge, after the inguinal surgical procedure, to 48 hours post-hospital discharge.

Primary Outcome Measurement Tool: Postoperative pain will be measured at three time the evening of the procedure, 24 hours post-discharge and 48 hours post-discharge) using the validated Parents Postoperative Pain Measure (PPPM) (See Appendix A).10 Pain scales will only be administered by parents once the patient has been discharged home. Patients usually recover from surgery for an average of two hours prior to being discharged from hospital.

Secondary Outcomes Measurement Tool: Secondary outcomes will be measured as follows: 1) Analgesic use postoperatively while still in the hospital. This will be recorded by a member of the care team on the patient's chart. Parents will record supplemental Tylenol administered in a standardized medication log for both arms of the study; 2) Frequency of emesis during recovery phase (in hospital and post discharge) recorded on patient case report form and recorded from the 48 hour phone call. 3) Time to discharge will be recorded from patient discharge sheet by research assistant 4) Adverse reactions (post discharge) will be recorded on patient case report form 5) Surgical complications (surgical site infection, bleeding, wound dehiscence) will be assessed by a physician or nurse practitioner at 6-8 week follow-up visit 6) First bowel movement post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric Patients between the ages of 10 months-5 years at presentation to clinic
2. Patients diagnosed with inguinal hernia or hydrocele, or undescended testes requiring surgical intervention by a trained physician
3. Patients requiring inguinal day surgery

Exclusion Criteria:

1. Patients who have undergone previous inguinal surgery
2. Patients with other co-morbidities
3. Patients unable to be prescribed Ibuprofen or Morphine
4. Chronic use of nonsteroidal anti-inflammatory drugs (NSAIDS) or opioids
5. Patients with renal or hepatic failure
6. Patients with coagulation disorders
7. Deviation to pre-established anesthesia protocol
8. Patients diagnosed with asthma or restrictive airways

Ages: 10 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Pain scales Post-Discharge from Hospital | Postoperative pain will be measured at three time the evening of the procedure, 24 hours post-discharge and 48 hours post-discharge) using the validated Parents Postoperative Pain Measure (PPPM)
  Assessed through validated and reliable Parents Postoperative Pain Measure (PPPM) by trained and blinded parent/guardian at 24 hours and at 48 hour following discharge from the hospital.

SECONDARY OUTCOMES:
Analgesic use post-operatively | Measured dosage post-surgery (on average 45 minutes later)
  Defined as the number of doses of Tylenol (15mg/kg) administered by PACU and SDSU nurses following surgery. Parents will record supplemental Tylenol administered in a pain diary for both arms of the study
Frequency of emesis (during hospital stay) | From the time surgical procedure is completed to discharge from the hospital. (Typically two to four hours)
  The frequency of emesis (vomiting) will be recorded by nurses at the recovery unit (post anesthetic care unit and same day surgery unit) during the patient's hospital stay.
Time to Discharge | Time from the end of the surgical procedure to discharge from hospital. (Typically two to four hours)
  The time it takes for the patient to be discharged from the hospital, beginning from when they first complete surgery.
Adverse reactions (during hospital stay) | Any complications that arise during the patient's recovery at the hospital (Typically two to four hours)
  Any complications that arise with the patient, during their recovery in the hospital.
Surgical complications | Surgical complications will be seen at the patient's 48-hour follow-up visit.
  Any surgical complications that arise during the patient's surgery (surgical site infection, bleeding, wound dehiscence) will be assessed by a physician or nurse practitioner at 48-will be seen by the physician or nurse practitioner at the patient's 48-hour follow-up visit.
First bowel movement post-surgery | The first bowel movement for the patient after surgery (Immediately after surgery to 3 Days post surgery)
  The first bowel movement post-surgery for the patient (during hospital stay or at home).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Braga, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada